CLINICAL TRIAL: NCT02860520
Title: Clinical Implication of the Molecular Diagnostic Retinitis Pigmentosa Molecular Diagnostic Using High Throughput Sequencing (RP-SEQ-HD)
Brief Title: Clinical Implication of Retinitis Pigmentosa Molecular Diagnostic Using High Throughput Sequencing.
Acronym: RP-SEQ-HD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5724
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa:
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The retinitis pigmentosa (RP) are genetic conditions that cause retinal degeneration leading to severe low vision and is the leading cause of consultation in reference centers dedicated to the ophthalmic genetics. These rare diseases are characterized by a triple heterogeneity (clinical, genetic and molecular), which made them unreachable by traditional molecular diagnostic sequencing technology by the large number of genes to be tested (> 190).

The advent of high-throughput sequencing (NGS) and targeted capture has opened unexpected possibilities of investigation and ultimately to improve the care of patients. This project aims to study the genetic and molecular epidemiology of an interregional french (grand EST) cohort of patients. Patients receive a detailed retinal phenotype (visual acuity, visual field, photographs of the fundus and ERG). Their DNA will be analyzed by NGS targets the 190 known genes (https://sph.uth.edu/retnet/).

This research will provide a molecular epidemiological cohort study compared to prior publications on the frequency of genes involved. The benefit for patients is important to: establish a mode of transmission of the disease and optimize genetic counseling (currently very empirical); establish phenotype-genotype correlations in the French population (very few studies to date) and from the data of international literature; identify patients likely to be included in future therapeutic protocols of research; identify patients with significant potential for future projects to identify new genes.

The primary purpose of the protocol is to use high throughput sequencing to identify pathogenic variants in genes involved in RP.

The secondary purposes will be the following:

* Determining the diagnostic yield
* Study the genotype-phenotype correlation.

The secondary purposes will be the following:

* Determining the diagnostic yield
* Study the genotype-phenotype correlation

ELIGIBILITY:
Inclusion Criteria:

* Subject of both sex, aged at least 2 years, being diagnosed with an RP, and/or having a family history of RP
* Informed about the results of the preliminary medical visit, or which (s) holder (s) parental authority or the guardian / curator has (have) was (been) informed
* Informed consent signed
* Affiliation to the French health system

Exclusion Criteria:

* The patient does not want to participate to the protocol
* Intercurrent diseases do not allow the practice of tests provided for this protocol
* Phenocopy
* Subject excluded or being excluded by another protocol
* Subject in emergency case
* Subject under judicial protection

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an RP and/or having a family history of RP
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-11-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a deleterious mutation | 18 months

SECONDARY OUTCOMES:
Percentage of positive diagnostic | 18 months
Number of gene with a genotype-phenotype correlation | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hélène DOLLFUS, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Service d'Ophtalmologie CHU Hôpital Général, Dijon
  - Service d'Ophtalmologie, Hôpital Robert Debré, CHR, Reims
  - Affections Rares en Génétique Ophtalmologique (CARGO) Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service d'Ophtalmologie, CHU BRABOIS, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No